CLINICAL TRIAL: NCT07363668
Title: Investigation of the Effects of Aromatherapy Foot Massage on Postoperative Pain, Sleep, and Recovery in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ümmügülsüm Dursun, Msc, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023/47
Record Dates: First submitted 2025-12-22; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2023-06

CONDITIONS: Cholelithiasis; Cholecystitis; Gallbladder Diseases; Postoperative Pain
Keywords: Nursing; Aromatherapy; Foot massage; Laparoscopic cholecystectomy; Sleep quality; Postoperative recovery
MeSH Terms: conditions — Cholelithiasis; Cholecystitis; Gallbladder Diseases; Pain, Postoperative; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy foot massage (Experimental): Patients receiving aromatherapy foot massage in addition to standard postoperative care
  Interventions: Other: aromatherapy foot massage
- control (No Intervention): Patients receiving standard postoperative care without aromatherapy massage

INTERVENTIONS:
Other: aromatherapy foot massage — Aromatherapy foot massage applied to both feet for 10 minutes approximately one hour after surgery and repeated six hours later.
  Arms: Aromatherapy foot massage

SUMMARY:
This randomized controlled study aims to evaluate the effects of aromatherapy foot massage on postoperative pain, sleep quality, and recovery in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
This study is a randomized controlled trial conducted in patients undergoing laparoscopic cholecystectomy. Eligible patients are randomly assigned to either an aromatherapy foot massage group or a control group receiving standard postoperative care.

In the intervention group, aromatherapy foot massage is applied to both feet for 10 minutes approximately one hour after surgery and repeated six hours later. The control group receives routine postoperative care without massage.

Pain intensity is assessed using the Visual Analog Scale (VAS). Sleep quality is assessed using the Visual Sleep Scale, and postoperative recovery is assessed using the Postoperative Recovery Index. Measurements are performed preoperatively and during the postoperative period according to the study protocol.

The study is conducted in accordance with ethical principles, and written informed consent is obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Patients undergoing laparoscopic cholecystectomy
* Able to communicate and provide informed consent
* Willing to participate in the study

Exclusion Criteria:

* Patients with cognitive impairment or communication difficulties
* Patients with chronic pain disorders
* Patients using continuous analgesic or sedative medication
* Patients with complications requiring intensive care
* Patients who decline to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
pain intensity (VAS score) | 5, 30, 60, 90, and 120 minutes after the massage session and on postoperative Day 1
  Pain intensity was assessed using the Visual Analog Scale (VAS), a 10-cm horizontal line ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain intensity.
postoperative recovery (postoperative recovery ındex score) | Baseline (preoperative) and postoperative Day 1
  Postoperative recovery was assessed using the Postoperative Recovery Index (PRI), a validated questionnaire used to evaluate patients' recovery after surgery. Higher scores indicate better postoperative recovery.

SECONDARY OUTCOMES:
sleep quality (visual sleep scale score) | Baseline (preoperative) and postoperative Day 1
  Sleep quality was assessed using the Visual Sleep Scale (VSS), a self-reported scale used to evaluate perceived sleep quality. Higher scores indicate better sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University Research and Application Center, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in an anonymized form upon request from researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From study completion
Access Criteria: •Who can access it: Authorized researchers and academic institutions. • Conditions: • Requesting researchers must obtain ethical committee approval from their institution. • Data will be shared in an anonymized form and for research purposes only. • Requests must be made in writing via PRS.